CLINICAL TRIAL: NCT03217318
Title: Reduction of Stent Associated Morbidity by Minimizing Stent Material: A Prospective Randomized Single-blind Study Assessing a Novel "Suture-Stent".
Brief Title: Reduction of Stent Associated Morbidity by Minimizing Stent Material.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Dominik Abt, Principal Investigator, Senior Physician Dept. of Urology, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTU 16.028 EKOS 17-00496
Record Dates: First submitted 2017-07-03; First posted 2017-07-14 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-02

CONDITIONS: Ureteral Stent Related Morbidity
Keywords: ureteral stent

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ureteral stenting with standard ureteral stent (Active Comparator): Group 1 will receive a standard ureteral stent. Diameter: 6F, length according to surgeons' estimation and patient's height.
  Interventions: Device: ureteral stenting with standard or modified ureteral stent
- ureteral stenting with suture-stent (Active Comparator): In Group 2, a modification of the standard ureteral stent will be inserted. The stent will be cut through obliquely according to the position of the ureteral calculus. The extend to be removed can be easily measured by the retrograde probing catheter and is replaced by a monofilament, non-absorbable suture as described previously by Vogt et al. (W J Urol, 2015). This suture can be easily attached by puncturing the bevelled stent end.
  Interventions: Device: ureteral stenting with standard or modified ureteral stent

INTERVENTIONS:
Device: ureteral stenting with standard or modified ureteral stent — Ureteral stenting because of kidney and or ureteral stones at the iliacal vessel crossing of the ureter or proximally

SUMMARY:
After providing informed consent, patients will be randomized into one of two groups (single-blinded): Group 1 will receive a standard Percuflex® (Boston scientific) ureteral stent. Diameter: 6F, length according to surgeons' estimation. Patients in Group 2 will receive a Suture-Stent adjusted to the individual stone location.

All participant receive standardized patient information, using a validated leaflet on ureteral stenting and associated morbidity.

In both groups, patients will complete the Ureteral Stent Symptoms Questionnaire (USSQ) 1 week after stent insertion, prior to stent removal (i.e. 2-6 weeks after insertion) and after (2-6 weeks) stent removal. USSQ results after stent removal serve as an assessment of "baseline symptoms". During secondary stone removal, stents are removed and ureteral dilatation / access is assessed.

The removed stents will be assessed for biofilm formation within the framework of an approved and ongoing study on the development of a Biofilm-model (EKSG 15/084). Potential complications and adverse events are assessed at all scheduled and unscheduled patient visits.

ELIGIBILITY:
Inclusion Criteria:

* Kidney stone(s) and/or ureteral stone(s) at the iliacal vessel crossing of the ureter or proximally
* Indication for ureteral stenting for the preparation of a secondary intervention
* Informed consent

Exclusion Criteria:

* Patients younger than 18 years
* Bilateral ureteral stenting
* Stenting because of malignant obstruction
* Mentally retarded patients
* Obstructive pyelonephritis at the time of stent insertion
* Additional operations performed during the stent indwelling time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Difference in Pain-Symptoms and Urinary-Symptoms as assessed by the validated questionnaire USSQ (ureteral stent symptoms questionnaire) between standard stent and Suture-Stent | One week after stent insertion and 2-6 weeks after removal
  Difference in the USSQ subscores ("Pain-Symptoms" and "Urinary-Symptoms") between standard stent and Suture-Stent (symptoms assessed one week after insertion and corrected for "baseline symptoms" by assessing symptom subscores 2-6 weeks after stent removal)

SECONDARY OUTCOMES:
Difference in Pain-Symptoms and Urinary-Symptoms as assessed by the validated questionnaire USSQ (ureteral stent symptoms questionnaire) between standard stent and Suture-Stent | 2-6 weeks after stent insertion and 2-6 weeks after removal
  Difference in the USSQ subscores ("Pain-Symptoms" and "Urinary-Symptoms") between standard stent and Suture-Stent (symptoms assessed before removal (i.e. 2-6 weeks after insertion) and corrected for "baseline symptoms" by assessing symptom subscores 2-6 weeks after stent removal).
Difference in total morbidity as assessed by the validated questionnaire USSQ (ureteral stent symptoms questionnaire) | 2-6 weeks after stent insertion and 2-6 weeks after removal
  Difference in the USSQ total score between standard ureteral stent and Suture- Stent (symptoms assessed before removal (i.e. 2-6 weeks after insertion) and corrected for "baseline symptoms" by assessing symptom subscores 2-6 weeks after stent removal).
Difference in type of morbidity as assessed by USSQ sub-scores and single-items (e.g. equal function, work incapacity, hematuria and others) between standard ureteral stent and Suture-Stent | 2-6 weeks after stent insertion and 2-6 weeks after removal
  Difference in the USSQ sub scores and items (i.e. general health, work performance, sexual matters, items, additional problems, GQ, assessment of haematuria: items U8 and U9) between standard ureteral stent and Suture-Stent (symptoms assessed before removal (i.e. 2-6 weeks after insertion) and corrected for "baseline symptoms" by assessing symptom subscores 2-6 weeks after stent removal).
Comparison of the ureteral expanse after stenting with the new Suture-Stent and the standard ureteral stent at the time of secondary intervention | 2-6 weeks after stent insertion
  Comparison of the ureteral expanse after stenting with the new Suture-Stent and the standard ureteral stent at the time of secondary intervention (measured by a retrograde ureterography) at three locations of the ureter (i.e. proximal, middle and distal ureter).
Differences of ureteral access with a 9.5 F ureterorenoscopy device after stenting with the new Suture-Stent or the standard ureteral stent at the time of secondary intervention (URS) | 2-6 weeks after stent insertion
  Differences of ureteral access with a 9.5 F ureterorenoscopy device after stenting with the new Suture-Stent or the standard ureteral stent at the time of secondary intervention (URS) measured by the success of: Entering the whole ureter or Insertion of an access sheath 14/12F; Complete stone removal.
Comparison of the mucosal irritation after stenting with the new Suture-Stent and the standard ureteral stent at the time of secondary intervention | 2-6 weeks after stent insertion
  Comparison of the mucosal irritation after stenting with the new Suture-Stent and the standard ureteral stent at the time of secondary intervention (measured by a grading: no, light, heavy irritation) at two locations (periostial and ureteral).
Comparison of practicability of Suture-Stent and standard ureteral stent | 2-6 weeks after stent insertion
  Comparison of practicability of Suture-Stent and standard ureteral stent (i.e. insertion time, problems with insertion or removal)
Comparison of the total biofilmmass and number of bacteria on stent surface between the Suture-Stent and standard ureteral stent | At the time of stent insertion and 2-6 weeks after insertion
  Comparison of the total biofilmmass and number of bacteria on stent surface between the Suture-Stent and standard ureteral stent measured at time of stent removal (2-6 weeks after insertion)
Microbiological investigation of the suture-part of the Suture-stent | 2-6 weeks after stent insertion
  Microbiological investigation of the suture-part of the Suture-stent: total biofilmmass, number of bacteria
Assessment of complications not assessed by USSQ during intervention and indwelling time (i.e. intraoperative complications, additional hospitalizations, prolongation of hospitalization, ureteral injuries) | At the time of stent insertion until 2-6 weeks after stent removal
  Assessment of complications not assessed by USSQ during intervention and indwelling time (e.g. perioperative adverse events according to Clavien-Dindo classification, stent dislocation or dysfunction during indwelling time).
Assessment of medication that had to be taken in both groups | At the time of stent insertion until 2-6 weeks after stent removal
  Assessment of medication that had to be taken in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Urological Department, Cantonal Hospital of St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No